CLINICAL TRIAL: NCT01255865
Title: Deep Tissue Thermometry 510(k) Premarket Notification Trial
Brief Title: Comparison Study of Core Temperature Thermometry Systems
Status: Completed | Type: Observational
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: Arizant 10-1026
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Thermometry Device Comparisons
Keywords: Thermometry; Deep Tissue Temperature; Core Temperature; Body Temperature; Rectal Temperature; Oral Temperature

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- A1 - up to 1 month: Age group 0 up to 1 month
- A2 - 1 to 3 months: Age group from 1 month to 3 months
- A3 - 3 months to 1 year: Age group from 3 months to 1 year
- B - 1 year to 5 years: Age group from older than 1y and younger than 5 years
- C - 5 years to 12 years: Age group from older than 5y and younger than 12 years
- D - 12 years to 21 years: Age group from older than 12 years and younger than 21 years
- E - 21 years and older: Age group older than 21 years

SUMMARY:
The purpose of this trial is the generation of clinical data required for a 510(k) submission to the FDA.

DETAILED DESCRIPTION:
The purpose of this trial is the generation of clinical data required for a 510(k) submission to the FDA. The trial design reflects elements desired by the FDA. The trial is designed to satisfy the relevant requirements of the FDA Guidance (March 1993) on the content of premarket notification [510(k)] submissions for clinical electronic thermometers and ISO/IEC 80601-2-56 Medical electrical equipment - Part 2-56: Particular requirements for basic safety and essential performance of clinical thermometers for body temperature measurement.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Subjects with skin disruptions on the forehead, dysautonomia, spinal cord injury, or taking barbiturates, thyroid preparations, antipsychotics, or who have had a recent (1wk) immunization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 120 subjects of any racial, gender, or ethnic background in who simultaneous measurments of deep tissue, oral, or rectal temperature can be made
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel i Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- See also: Outcomes Research Consortium — http://www.or.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Age 1: Age group 0 up to 1 month
- Age 2: Age group from 1 month to 3 months
- Age 3: Age group from 3 months to 1 year
- Age 4: Age group from older than 1y and younger than 5 years
- Age 5: Age group from older than 5y and younger than 12 years
- Age 6: Age group from older than 12 years and younger than 21 years
- Age 7: Age group older than 21 years
Period: Overall Study
Arm/Group | Age 1 | Age 2 | Age 3 | Age 4 | Age 5 | Age 6 | Age 7
Started | 1 | 10 | 10 | 30 | 20 | 20 | 20
Completed | 1 | 10 | 10 | 30 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age1: Age group 0 up to 1 month
- Age2: Age group from 1 month to 3 months
- Age3: Age group from 3 months to 1 year
- Age4: Age group from older than 1y and younger than 5 years
- Age5: Age group from older than 5y and younger than 12 years
- Age6: Age group from older than 12 years and younger than 21 years
- Age7: Age group older than 21 years
- Total: Total of all reporting groups
Arm/Group | Age1 | Age2 | Age3 | Age4 | Age5 | Age6 | Age7 | Total
Number analyzed (Participants) | 1 | 10 | 10 | 30 | 20 | 20 | 20 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 10 | 10 | 30 | 20 | 20 | 0 | 91
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Subjects were categorized by age group but actual age was not collected. | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected | NA (NA) — Subjects were categorized by age group but actual age was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 10 | 14 | 9 | 12 | 50
  Male | 1 | 7 | 8 | 20 | 6 | 11 | 8 | 61
Region of Enrollment [Number; unit: participants]
  United States | 1 | 10 | 10 | 30 | 20 | 20 | 20 | 111

OUTCOME MEASURES:

1. Primary Outcome: Temperature Agreement in Degrees Celsius.
Description: Temperature Agreement/Bias (Zero heat flux thermometry temperature minus oral or rectal temperature) between simultaneously-acquired oral or rectal and forehead deep tissue temperatures.
Time Frame: Upon enrollment
Measure: Mean (Standard Deviation); unit: Temperature in Celsius
Arm/Group | Age1 | Age2 | Age3 | Age4 | Age5 | Age6 | Age7
Number analyzed (Participants) | 1 | 10 | 10 | 30 | 20 | 20 | 20
Temperature in Celsius | NA (NA) — Only a single subject in this group so mean and SD at not calculated | 0.5 (0.59) | 0.5 (0.47) | 0.4 (0.43) | 0.5 (0.32) | 0.3 (0.47) | 0.0 (0.02)

ADVERSE EVENTS:
Time Frame: Immediately upon enrollment
Arm/Group | Age1 | Age2 | Age3 | Age4 | Age5 | Age6 | Age7
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/10 | 0/10 | 0/30 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/10 | 0/10 | 0/30 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/1 | 0/10 | 0/10 | 0/30 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No